CLINICAL TRIAL: NCT04702906
Title: Trimetazidine As a Potential Adjuvant Therapy in Acute Aluminum Phosphide Poisoning-induced Cardiotoxicity: A Randomized Controlled Clinical Trial
Brief Title: Trimetazidine As a Potential Adjuvant Therapy in Acute Aluminum Phosphide Poisoning-induced Cardiotoxicity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nadia Helal, lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aluminum Phosphide Poisoning
Record Dates: First submitted 2020-12-15; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Aluminum Phosphide Poisoning
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): All patients will continue to receive the standard treatment, which is determined by the attending physician who maintains clinical responsibility for all patients. Conventional standard treatment included using inotropes, fluids and electrolytes resuscitation, intubation, mechanical ventilation, and antiarrhythmic agents if indicated.
  Interventions: Other: standard treatment
- trimetazidine group (Active Comparator): The trimetazidine group will receive conventional standard treatment plus Trimetazidine dihydrochloride "metacardia" ® (20 mg three times daily produced by Pharco-Egypt) will be administered twice every 24 hours until at least treatment is no longer needed.
  Interventions: Other: standard treatment; Drug: trimetazidine hydrochloride "metacardia" ® 20 mg tablet

INTERVENTIONS:
Other: standard treatment — Standard treatment if indicated.
Drug: trimetazidine hydrochloride "metacardia" ® 20 mg tablet — trimetazidine hydrochloride "metacardia" ® (20 mg three times daily produced by Global NAPI Pharmaceuticals-Egypt)
  Arms: trimetazidine group

SUMMARY:
The aim of the present study is to evaluate the potential adjuvant therapeutic effect of trimetazidine in treatment of acute AlP poisoning-induced cardiotoxicity.

DETAILED DESCRIPTION:
Aluminium phosphide (AlP) is an inorganic phosphide. It is used as a fumigant to protect stored grains from insects, rodents and other pests.It is a solid fumigant widely used in Egypt as a grain preservative. Its tablets are commonly used due to their low cost, high efficacy, and availability .

Toxic effects of AlP are related to phosphine gas release when AlP comes in contact with moisture or gastric acidity. Phosphine gas is rapidly absorbed from the gastrointestinal tract and lungs inhibiting cytochrome-c oxidase and oxidative phosphorylation which results in adenosine triphosphate depletion and resulting cellualr death.

The direct toxic effects of phosphine on cardiac myocytes, fluid loss and adrenal gland can induce profound circulatory collapse. Phosphides and phosphine can exert a direct corrosive effect on body tissues.

Toxic manifestations usually appear rapidly upon phosphide exposure. Impaired myocardial contractility, fluid loss, pulmonary edema, metabolic acidosis and acute renal failure are the most frequent manifestations. Disseminated intravascular coagulation and hepatic necrosis may also occur. Patients generally die due to multi-organ failure .However, myocardial damage- induced cardiovascular collapse is reported to be the primary cause of death.

Severity of manifestations depends on different factors such as dose, exposure route, and time delay before treatment initiation. Diagnosis is based on history of exposure, garlic odor of the breath, suggestive clinical manifestations and detection of phosphine gas in gastric aspirate or breath.

Treatment of acute AlP toxicity is mainly supportive as there is no specific antidote since the exact mechanism of toxicity is still unknown. The most important factor is resuscitation of shock. Many researches are directed towards finding a specific treatment for this fatal poison.

Trimetadizine is described as the first cytoprotective anti-ischemic agent developed. It has a protective of the myocardium due to its preservation of oxidative metabolism. It improves myocardial glucose utilization through inhibition of long-chain 3-ketoacyl CoA thiolase activity, which results in a reduction in fatty acid oxidation and a stimulation of glucose oxidation .

Trimetadizine reduces the tissue accumulation of malonyldialdehyde, the lipid peroxidation index, and the sodium influx related to activation of the Na+ -K + pump. Moreover, it lack of haemodynamic effects. These effects result in a decrease in the cellular accumulation of calcium and improved intracellular ATP levels).

Oral administration of the anti-ischaemic drug trimetazidine, was tried in a case report of occupational inhalation exposure to phosphine gas from AlP. It was temporally associated with clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this study will be diagnosed as acute aluminum phosphide poisoning by history and clinical pictures.

  * Age is18 years or older.

Exclusion Criteria:

* Pregnant and lactating women.
* Patients with ingestion or exposure to other substances in addition to aluminum phosphide.
* Patients with other major medical conditions (e.g. cardiovascular disease, diabetes mellitus, renal or hepatic failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Mortality | 7 days
  mortality rate

SECONDARY OUTCOMES:
Duration of ventilation | 7 days
  Duration of mechanical ventilation